CLINICAL TRIAL: NCT05017987
Title: A Phase I Clinical Trial to Compare and Evaluate Safety and Pharmacokinetic Characteristics After Administration of ATB-101 or Co-administration of ATB-1011 and ATB-1012 in Healthy Adult Volunteers
Brief Title: Clinical Trial to Compare Pharmacokinetics After Administration of ATB-101 or Co-administration of ATB-1011 and ATB-1012
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Autotelicbio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ATB-101-002
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Healthy Adult Volunteers

STUDY DESIGN:
Intervention Model Description: Open, Randomization, single oral administration, 2 Intervention group, crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A=Reference-Test (Active Comparator): T(Test drug): ATB-101 R1(Reference drug1): ATB-1011 R2(Reference drug2): ATB-1012
  First stage: co-administration of R1 and R2, single dose and then Washout: 7days and then Second stage: administration of T, single dose
  Interventions: Drug: ATB-101, ATB-1011, ATB-1012
- Sequence B=Test-Reference (Active Comparator): First stage: administration of T, single dose and then Washout: 7days and then Second stage: co-administration of R1 and R2, single dose
  Interventions: Drug: ATB-101, ATB-1011, ATB-1012

INTERVENTIONS:
Drug: ATB-101, ATB-1011, ATB-1012 — 1. Test drug
     - Code name: ATB-101
  2. Control drug1
     * Code name: ATB-1011
     * Active ingredient: Olmesartan
  3. Control drug2
     * Code name: ATB-1012
     * Active ingredient: Dapagliflozin
  Other Names: ATB-1011 brand name: Olmetec; ATB-1012 brand name: Forxiga

SUMMARY:
To compare and evaluate safety and pharmacokinetic Characteristics after administration of ATB-101 or co-administration of ATB-1011 and ATB-1012 in fasted Healthy Adult Volunteers

DETAILED DESCRIPTION:
Pharmacokinetic endpoints

1. Primary endpoint : AUCt, Cmax of Dapagliflozin, Olmesartan
2. Secondary endpoint : AUC∞, Tmax, t1/2, CL/F, Vd/F of Dapagliflozin, Olmesartan

Safety evaluation

1. Adverse reactions (but only in case of TEAE)
2. Concomitant drugs
3. Vital signs
4. Laboratory test

ELIGIBILITY:
Inclusion Criteria:

* Those who are over 19 years old at the screening visit
* Those who do not have clinically significant congenital or chronic diseases and have no pathological symptoms or findings upon medical examination at the screening visit
* Those who determined as suitable study subjects by the principal investigator
* A person who signs the consent form at will, after hearing and understanding a sufficient explanation of the purpose, contents, characteristics of the investigational product, and expected adverse reactions of this clinical trial

Exclusion Criteria:

* Those who have a clinically significant disease or have a history of such disease
* Those who have a history of gastrointestinal surgery
* Those who have taken drugs that induce and inhibit metabolism enzymes such as barbital drugs
* Those who participated in other clinical trials or bioequivalence studies and administered the investigational products within 6 months of the first administration date.
* Those who donated whole blood within 2 months or donated components within 2 weeks, or received a blood transfusion within 1 month of the first administration date

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-06-19 (Actual); Primary Completion 2021-07-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
AUCt of Olmesartan | Day1(first stage), Day8(scond stage)
  Area under the concentration-time curve
Cmax of Olmesartan | Day1(first stage), Day8(scond stage)
  Maximum concentration of drug in plasma
AUCt of Dapagliflozin | Day1(first stage), Day8(scond stage)
  Area under the concentration-time curve
Cmax of Dapagliflozin | Day1(first stage), Day8(scond stage)
  Maximum concentration of drug in plasma

SECONDARY OUTCOMES:
AUC∞ of Olmesartan | Day1(first stage), Day8(scond stage)
  Area under the plasma drug concentration-time curve from time 0 to infinity
Tmax of Olmesartan | Day1(first stage), Day8(scond stage)
  Time to maximum plasma concentration
T1/2 of Olmesartan | Day1(first stage), Day8(scond stage)
  Terminal elimination half-life
CL/F of Olmesartan | Day1(first stage), Day8(scond stage)
  Apparent total clearance of the drug from plasma after oral administration
Vd/F of Olmesartan | Day1(first stage), Day8(scond stage)
  Apparent volume of distribution after non-intravenous administration
AUC∞ of Dapagliflozin | Day1(first stage), Day8(scond stage)
  Area under the plasma drug concentration-time curve from time 0 to infinity
Tmax of Dapagliflozin | Day1(first stage), Day8(scond stage)
  Time to maximum plasma concentration
T1/2 of Dapagliflozin | Day1(first stage), Day8(scond stage)
  Terminal elimination half-life
CL/F of Dapagliflozin | Day1(first stage), Day8(scond stage)
  Apparent total clearance of the drug from plasma after oral administration
Vd/F of Dapagliflozin | Day1(first stage), Day8(scond stage)
  Apparent volume of distribution after non-intravenous administration

CONTACTS AND LOCATIONS:
Overall Officials: Jaewoo Kim, Principal Investigator — H + Yangji Hospital
Locations (1):
- H Plus Yangji Hospital, Seoul, Gwanak-gu, South Korea

IPD SHARING:
Plan to Share IPD: No